CLINICAL TRIAL: NCT00250991
Title: Combined Approach to Lysis Utilizing Eptifibatide and rt-PA in Acute Ischemic Stroke (CLEAR Stroke) Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Arthur Pancioli, MD, University of Cincinnati College of Medicine, Department of Emergency Medicine
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: P50NS044283 (NIH)
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Stroke
Keywords: stroke; integrilin; eptifibatide; activase; recombinant tissue plasminogen activator; rt-PA; recombinant t-PA; SPOTRIAS
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator; Eptifibatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: activase
Drug: integrilin

SUMMARY:
The purpose of this study is determine the effects of using of a combination of two drugs--integrilin (eptifibatide) and activase (recombinant tissue plasminogen activator, rt-PA, or recombinant t-PA)--to dissolve blood clots in patients who have a stroke.

DETAILED DESCRIPTION:
The Combined Approach to Lysis Utilizing Eptifibatide and rt-PA in Acute Ischemic Stroke (CLEAR Stroke) trial is part of the Specialized Program on Translational Research in Acute Stroke (SPOTRIAS). The overall goals of SPOTRIAS are to enhance delivery of acute stroke patient care and train acute stroke translational researchers.

Stroke most often occurs when blood flow to the brain stops because it is blocked by a blood clot. When a blood clot blocks the blood supply to the brain, parts of the brain may not get enough blood and oxygen to survive. As a result, permanent brain damage can occur, which can affect a person's ability to walk, talk, and function independently. In order to reduce the risk of permanent damage, it is important to restore blood flow to the brain as quickly as possible.

The CLEAR Stroke study will enroll 100 participants with acute stroke due to a blood clot. The purpose of this multi-center, randomized, double-blind study is to determine the effects of using a combination of two drugs, integrilin (or eptifibatide) and activase (or recombinant tissue plasminogen activator, rt-PA, recombinant t-PA), to dissolve blood clots. More specifically, the CLEAR study is being done to determine if a lower dose of activase, given in combination with a second drug, integrilin, is a safe treatment for acute stroke.

Activase, used alone, is already approved by the Food and Drug Administration (FDA) as treatment for patients with a stroke caused by blockage of an artery in the brain and when given within 3 hours of the onset of stroke symptoms. Integrilin is also already FDA-approved as a treatment for blood clots causing heart attack. The investigational aspect of this study is the use of integrilin for a stroke victim in combination with activase.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a serious measurable neurological deficit on the NIH Stroke Scale due to focal brain ischemia.
* An NIH Stroke Scale score >5 at the time that intravenous study drug is begun.
* Age: 18 through 80 years (i.e. candidates must have had their 18th birthday, but not had their 81st birthday).
* Intravenous therapy must be initiated within 3 hours of onset of stroke symptoms.

Exclusion Criteria:

* History of stroke in the past 3 months.
* Previous intra-cranial hemorrhage, neoplasm, subarachnoid hemorrhage, or arterial venous malformation
* Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT scan is normal
* Hypertension at time of treatment; systolic BP > 185 or diastolic > 110 mmHg or aggressive measures to lower blood pressure to below these limits are needed.
* Presumed septic embolus
* Presumed pericarditis including pericarditis after acute myocardial infarction
* Recent (within 30 days) surgery or biopsy of parenchymal organ
* Recent (within 30 days) trauma, with internal injuries or ulcerative wounds
* Recent (within 90 days) severe head trauma or head trauma with loss of consciousness
* Any active or recent (within 30 days) serious systemic hemorrhage
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; or oral anticoagulant therapy with prothrombin time greater than 15 or INR > 1.4
* Baseline lab values: positive urine pregnancy test, glucose < 50 or > 400 mg/dl, platelets <100,000 /mm3, Hct <25 %, or creatinine > 4 mg/dl
* Ongoing renal dialysis, regardless of creatinine
* If heparin has been administered within 48 hours, the patient must have a normal partial thromboplastin time (PTT)
* Arterial puncture at a non-compressible site or a lumbar puncture in the previous 7 days
* Seizure at onset of stroke
* Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations
* Other serious, advanced, or terminal illness or any other condition that the investigator feels would pose a significant hazard to the patient if rt-PA or eptifibatide therapy were initiated
* Patients whose peripheral venous access is so poor that they are unable to have two standard peripheral Intravenous lines started.
* Current participation in another research drug treatment protocol. Patient cannot start another experimental agent until after 90 days
* Informed consent is not or cannot be obtained
* Any known history of amyloid angiopathy.

Exclusion Criteria/CT Scan:

* High density lesion consistent with hemorrhage of any degree.
* Significant mass effect with midline shift.
* Large (more than 1/3 of the middle cerebral artery) regions of clear hypodensity on the baseline CT scan. Sulcal effacement and/or loss of grey-white differentiation alone are not contraindications for treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2003-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint in this safety study will be the incidence of symptomatic intracranial hemorrhage . | within 36 hours
The primary measure of early beneficial drug activity will be the incidence of early neurological improvement, as measured by the NIHSSS </= 2 | at 24 hours from symptom onset

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Pancioli, MD, Principal Investigator — University of Cincinnati College of Medicine, Department of Emergency Medicine
Locations (19):
- United States (19):
  - Barrow Neurologic Institute, St. Joseph's Hospital and Medical Center, 350 West Thomas Rd, Phoenix, Arizona
  - University of California, Los Angeles, UCLA Medical Center, 10833 Le Conte Ave., Los Angeles, California
  - Santa Monica-UCLA Medical Center, 1250 16th Street, Santa Monica, California
  - St. John's Health Center, 1328 22nd St, Santa Monica, California
  - St. Elizabeth Medical Center South, One Medical Village Drive, Edgewood, Kentucky
  - Jewish Hospital Louisville, Jewish Hospital Healthcare Services Inc., 200 Abraham Flexner Way, Louisville, Kentucky
  - University of Michigan, University of Michigan Health System, 1500 E. Medical Center Drive, TC B1354, Box 0303, Ann Arbor, Michigan
  - Long Island Jewish, North Shore-Long Island Jewish Health System, 270-05 76 Avenue, New Hyde Park, New York
  - The Christ Hospital, 2139 Auburn Ave., Cincinnati, Ohio
  - University of Cincinnati, University Hospital, 234 Goodman Ave., Cincinnati, Ohio
  - Good Samaritan Hospital, 375 Dixmyth Ave.,, Cincinnati, Ohio
  - The Jewish Hospital of Cincinnati, 4777 East Galbraith Rd,, Cincinnati, Ohio
  - Mercy Hospital, Western Hills, 3131 Queen City Ave., Cincinnati, Ohio
  - Mercy Hospital, Mt Airy, 2446 Kipling Ave., Cincinnati, Ohio
  - Bethesda North Hospital, 10500 Montgomery Rd, Montgomery, Ohio
  - Lehigh Valley Hospital, 1200 South Cedar Crest Blvd, Allentown, Pennsylvania
  - University of Pennsylvania, University of Pennsylvania Medical Center, 3400 Spruce Street, Philadelphia, Pennsylvania
  - Brown University, Rhode Island Hospital, 593 Eddy St., Providence, Rhode Island
  - Vanderbilt University, University Hospital, 1211 22nd Ave. S., Nashville, Tennessee